CLINICAL TRIAL: NCT06732544
Title: Effect of Multisensory (Snoezelen) Environment on Birth Outcomes, Newborn Health Parameters and Birth Memory: Randomized Controlled Study
Brief Title: Effect of Multisensory (Snoezelen) Environment on Birth Outcomes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Collaborators: Ege University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AU_Eliftez
Record Dates: First submitted 2024-05-25; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Healthy
Keywords: birth enviroment; newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experiment group (Experimental): These women will spend labor in the snoezelen room.
  Interventions: Other: snoezelen room
- control group (Other): These women will spend the duration of labor in a standard delivery room.
  Interventions: Other: routine delivery room

INTERVENTIONS:
Other: snoezelen room — During the travail, projectors, starry ceiling visuals and blue light LEDs will be used for visual stimuli, speakers will be used as auditory stimuli, diffusers will be used for olfactory stimuli, and therapy dough will be used for touch stimuli.
  Arms: experiment group
Other: routine delivery room — General practice
  Arms: control group

SUMMARY:
Giving birth is a fundamental life event that women will remember throughout their lives. While seeking perfection for the birth environment, much can be learned from other areas of expertise and different pursuits can be undertaken. An example of this is "Snoezelen rooms". In the Snoezelen environment, it is aimed to relax the woman by stimulating various senses, including visual and auditory, and by diverting attention. The room design is a combination of light music, aquarium, optical illusions and aromatic oils. This study will be conducted in a randomized controlled manner to examine the effects of a multi-sensory (snoezelen) environment on birth outcomes, newborn health parameters and birth memory.

ELIGIBILITY:
Inclusion Criteria:

* Those who are between the ages of 18-35
* Having a singleton pregnancy between 38-42 weeks of pregnancy
* Primiparous
* Labor started spontaneously
* In the latent phase of labor
* Without uterine contraction anomaly
* The leading part of the fetus is the head (in vertex position)
* No analgesia was applied
* There is no indication for cesarean section
* Amniotomy is not performed
* Fetal weight over 2500 g, fetal weight not over 4000 gr
* Pregnant women who do not have communication problems will be included in the study.

Exclusion Criteria:

* Reporting hearing, vision, smell and balance problems
* Allergy, asthma, COPD, migraine, vertigo, epilepsy, etc.
* Declaring that they have a chronic disease
* Declaring that they have a psychiatric history or a diagnosed psychological disorder
* Declaring that they have a risky health condition related to pregnancy (preeclampsia, gestational DM, etc.),
* Those who report smoking, alcohol and/or substance use
* Reports that he/she has sensory sensitivity
* Declaring an allergy to lavender (Lavandula angustifolia Mill.) or lavender oil
* Declaring that there is a person with special needs in the family
* Participated in the study voluntarily and then gave up
* Pregnant women who develop any possible side effects during the study will not be included in the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnancy women
Enrollment: 23 (Estimated)
Dates: Start 2024-09-08 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Personal information form | on admission to the hospital
  With this form, developed by the researcher taking into account literature knowledge, data on women's demographic information such as age, education level, and obstetric characteristics such as whether the pregnancy is planned and the current gestational week will be obtained (Hauck et al., 2008; Manesh et al. 2015).
birth follow-up form | at the beginning of the third stage of childbirth
  With the follow-up form prepared to evaluate the birth process using the literature, the duration of the stages during labor and the synthetic oxytocin status used will be evaluated. While these practices are evaluated, the researcher will be present in the environment only as an observer, and the practices determined as a result of the observation will be noted on the Birth Monitoring Form (Olcese et al., 2013 Momeni et al., 2020).
Birth Memory and Recall Scale | 24 hours after birth
  In order to evaluate women's postpartum birth memories, their birth memories, and their experiences regarding birth memories, DHHÖ conducted a study by Foley et al. (2014). It was adapted into Turkish by Topkara & Çağan (2021).

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya University Hospital, Amasya, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the article was published